CLINICAL TRIAL: NCT06748092
Title: Clinical Validation of iCare IC1000 Tonometer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TA032-135
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Masking Description: Investigator cannot see the measurement results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- iCare IC1000 vs GAT, iCare IC200 and Perkins (Experimental)
  Interventions: Device: iCare IC1000; Device: iCare IC200; Device: GAT; Device: Perkins

INTERVENTIONS:
Device: iCare IC1000 — Measurement of Intraocular Pressure (IOP) in sitting and supine position
Device: iCare IC200 — Measurement of Intraocular Pressure (IOP) in sitting and supine position
Device: GAT — Measurement of Intraocular Pressure (IOP) in sitting position
Device: Perkins — Measurement of Intraocular Pressure (IOP) in supine position

SUMMARY:
Clinical validation of iCare IC1000 tonometer per ANSI Z80.10:2014 standard

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Exclusion Criteria:

* Subjects with only one functional eye
* Subjects having poor or eccentric fixation in the study eye
* High corneal astigmatism >3D in the study eye
* Central corneal scarring
* History of prior incisional glaucoma surgery or corneal surgery, including corneal refractive laser surgery in the study eye
* Microphthalmos
* Buphthalmos
* Contact lens use within one week of continuous wear and within one hour if lens is worn occasionally
* Dry eyes (clinically significant)
* Lid squeezers - blepharospasm
* Nystagmus
* Keratoconus
* Any other corneal or conjunctival pathology or infection relevant to this study
* Central corneal thickness greater than 600 µm or less than 500 µm in the study eye
* Cataract Extraction within last 2 months in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Demonstrate compliance with ANSI Z80.10:2014-Ophthalmics-Ophthalmic Instruments-Tonometers | Through study completion, an average of 6 months
  Subjects will be distributed into Low IOP, Medium IOP, and High IOP groups based on the reference tonometer measurements. The iCare IC1000 Tonometer measurements shall be within +/-5.0 mmHg of the reference tonometer measurements in all groups.

SECONDARY OUTCOMES:
Retrospective analysis of "Quick Measure" mode | Through study completion, an average of 6 months
  The secondary objective of this study is to do a retrospective analysis of "Quick Measure" mode. Instead of 6 shots that are taken in Default Measure, Quick Measure takes only 2 shots (or 3 shots if the difference between the first two shots is greater than 2 mmHg). The Quick Measure results are calculated retrospectively from the raw data of the Default Measure results. Quick Measure comparison to reference measurements is done similarly as with Default Measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health/Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No